CLINICAL TRIAL: NCT01330277
Title: Biomarkers for Hunter Syndrome: An International, Multicenter, Observational, Longitudinal Protocol
Brief Title: Biomarkers for Hunter Syndrome
Acronym: BioHunter
Status: Terminated | Type: Observational
Why Stopped: Study no longer pursued.
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BH 06-2018
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Hunter Syndrome; Mucopolysaccharidosis II; Hunter's Syndrome, Mild Form; Hunter's Canal Syndrome
Keywords: Hunter Disease; Biomarker
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample applied on the Dry Blood Spot (DBS) Filtercard (Centocard®)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Hunter syndrome: Participants diagnosed with Hunter syndrome (Mucopolisaccharidosis type 2) aged between 2 months to 50 years

SUMMARY:
International, multicenter, observational, longitudinal study to establish Hunter Syndrom biomarker/s and to explore the clinical robustness, specificity, and long-term variability of these biomarker/s

DETAILED DESCRIPTION:
Mucopolysaccharides are long chains of sugar carbohydrates, found within the cells that help build bone, cartilage, tendons, cornea, skin, and connective tissue. Glycosaminoglycans (GAGs) are also found in the fluids that lubricate joints. Mucopolysaccharidosis (MPS) are part of the Lysosomal Storage Disorder (LSD) family, a group of more than 40 genetic diseases, and occur when a particular enzyme exists in a small quantity or is missing altogether. The effect is the accumulation of GAGs in the cells, blood, and connective tissues, resulting in permanent and progressive cellular damage which affects appearance, physical abilities, organ and system functioning and, in most cases, mental development.

MPS2 (also called Hunter syndrome) is a hereditary, progressive, multisystemic disorder, caused by mutations in the IDS gene coding for the enzyme iduronate sulfatase (Ids). It is the only type of mucopolysaccharidosis that is X-linked, therefore, if mothers are carriers, there is a 50 percent chance for males to be born with the disease.

MPS2 has a wide range of symptoms that vary in severity, which can be managed with enzyme replacement therapy (ERT). ERT is unable to cross the blood-brain barrier, therefore it addresses strictly extra-neurological manifestations. On this note, further efforts are being made to develop novel therapies, in the attempt to stop the disease progression and to offer a better quality of life to the patients.

As MPS2 is very rare and many medical professionals only see a few or no patients in their lifelong practice, genetic testing is crucial for diagnosis. This study thrives to identify, validate, and monitor potential biomarker/s for MPS2 in genetically confirmed samples.

ELIGIBILITY:
INCLUSION CRITERIA:

* Male individuals
* Informed consent is obtained from the participant's parent/legal guardian
* The participant is aged between 2 months and 50 years of age
* The diagnosis of MPS II is genetically confirmed by CENTOGENE

EXCLUSION CRITERIA:

* Females
* Informed consent is not provided by the participant's parent/legal guardian
* The participant is younger than 2 months or older than 50 years of age
* The diagnosis of MPS II is not genetically confirmed by CENTOGENE

Ages: 2 Months to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Male
Study Population: Male participants with genetically confirmed Hunter syndrome (Mucopolisaccharidosis type 2 or MPS2)
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Identifying MPS II biomarkers | 36 weeks
  All samples will be analyzed for the identification of biomarker/s via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS) and compared to merged control, in order to establish the disease-specific biomarker/s. The LC/MRM-MS is performed on an ABSciex 6500 triple quadrupole mass spectrometer, coupled with a Waters Acquity UPLC.

SECONDARY OUTCOMES:
To explore the clinical robustness, specificity, and long-term variability of MPS II biomarkers | 36 months
  Samples will be analyzed for the identified biomarker candidates via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS) and compared to merged control, in order to establish the disease-specific biomarker/s. The LC/MRM-MS is performed on an ABSciex 6500 triple quadrupole mass spectrometer, coupled with a Waters Acquity UPLC.

CONTACTS AND LOCATIONS:
Overall Officials: Arndt Rolfs, Prof. Dr., Principal Investigator — CENTOGENE GmbH Rostock
Locations (4):
- Mexico (4):
  - Private Practice, Cancún, Quintana Roo
  - Hospital Pediatrico de Sinaloa, Culiacán, Sinaloa
  - Centenario Hospital Miguel Hidalgo, Aguascalientes
  - Hospital Infantil de Tampaulipas, Ciudad Victoria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: CENTOGENE is a rare disease company focused on transforming clinical, genetic, and biochemical data into medical solutions for patients. — https://www.centogene.com/